CLINICAL TRIAL: NCT00789451
Title: The Effect of Ischaemic-reperfusion on the Endogenous Fibrinolysis in Man
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Aarhus (Other); University of Oxford (Other)
Responsible Party: Christian M Pedersen, clinical research fellow, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CMP 1
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Ischaemic Heart Diseases
Keywords: Ischaemia reperfusion; t-PA; Fibrinolysis; Endothelial function
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Sham Comparator): no ischaemia - only sham. Blood pressure cuff inflation up till 10 mmHg on the upper arm for 20 mins.
  Interventions: Procedure: Forearm vascular study
- 2 (Active Comparator): Ischaemia 20 minutes. Blood pressure cuff will be inflated around the upper arm for 20 minutes to induce ischaemia.
  Interventions: Procedure: Forearm vascular study

INTERVENTIONS:
Procedure: Forearm vascular study — Forearm blood flow measured by venous occlusion plethysmography during interarterial infusion of substance P (2,4,8 pmol/min). Venous blood sampling via cannula in antecubital fossa.

SUMMARY:
Heart attacks are usually caused by a blood clot blocking an artery supplying blood to the heart. Current treatments are designed at relieving this blockage as quickly as possible to minimise damage to the heart muscle. However in restoring the supply of blood local damage known as "ischaemia-reperfusion injury" may occur. The aim of this study is to assess how clot forming and clot dissolving pathways are affected during this process, and examine the role of a natural inflammatory hormone, bradykinin. This will help us to understand the mechanism by which ischaemia-reperfusion injury may occur and to devise new treatments for heart attacks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18-65 years of ages, non-smokers.

Exclusion Criteria:

* Any concurrent illness or chronic medical condition. Concurrent use of vasoactive medication. Smoking history.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Net t-PA release from the endothelium after ischaemia reperfusion | Throughout the study

SECONDARY OUTCOMES:
Change in forearm blood flow after ischaemia reperfusion | throughout the study
Change in platelet-monocyte-binding after ischaemia reperfusion | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD, FRCP, Study Director — University of Edinburgh; Rajesh K Kharbanda, PhD, FRCP, Study Director — University of Oxford
Locations (1):
- University of Edinburgh, 49 Little France Crescent, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Pedersen CM, Cruden NL, Schmidt MR, Lau C, Botker HE, Kharbanda RK, Newby DE. Remote ischemic preconditioning prevents systemic platelet activation associated with ischemia-reperfusion injury in humans. J Thromb Haemost. 2011 Feb;9(2):404-7. doi: 10.1111/j.1538-7836.2010.04142.x. No abstract available. PMID 21083644